CLINICAL TRIAL: NCT04024202
Title: The DRAIHA Study: Data Registry of AutoImmune Hemolytic Anemia, to Improve Diagnostic Testing for the Development of Personalized Treatment Protocols in AIHA Patients
Brief Title: Data Registry of Auto Immune Hemolytic Anemia
Acronym: DRAIHA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sanquin Research & Blood Bank Divisions (Other)
Collaborators: Leiden University Medical Center (Other); Radboud University Medical Center (Other); UMC Utrecht (Other); Maastricht University Medical Center (Other); Erasmus Medical Center (Other); Haga Hospital (Other); Isala (Other); Jeroen Bosch Ziekenhuis (Other); St. Antonius Hospital (Other); Onze Lieve Vrouwe Gasthuis (Other); Spaarne Gasthuis (Other); Amsterdam University Medical Center (Other); Prothya Biosolutions (Industry)
Responsible Party: Sponsor
Other Study IDs: PPOC 15-27
Record Dates: First submitted 2019-05-31; First posted 2019-07-18 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Autoimmune Hemolytic Anemia
MeSH Terms: conditions — Anemia, Hemolytic, Autoimmune

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples from patients (older than 16 years) and blood donors (older than 18 years) and urine samples from the first 20 included patients in each of the participating hospitals, will be collected for experimental diagnostic testing at inclusion (T0) and after 1-1,5 year (T1) of follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: 1. Patients with a positive DAT, a positive eluate and signs of hemolysis
  2. Patients with a positive DAT with complement only, negative eluate, but with hemolysis
- Blood donors: Blood donors with a positive direct antiglobulin test and a positive eluate and/or clinically relevant cold auto-antibodies

SUMMARY:
In autoimmune hemolytic anemia (AIHA) auto-antibodies directed against red blood cells (RBCs) lead to increased RBC clearance (hemolysis). This can result in a potentially life-threatening anemia. AIHA is a rare disease with an incidence of 1-3 per 100,000 individuals. An unsolved difficulty in diagnosis of AIHA is the laboratory test accuracy. The current 'golden standard' for AIHA is the direct antiglobulin test (DAT). The DAT detects autoantibody- and/or complement-opsonized RBCs. The DAT has insufficient test characteristics since it remains falsely negative in approximate 5-10% of patients with AIHA, whereas a falsely positive DAT can be found in 8% of hospitalized individuals. Also apparently healthy blood donors can have a positive DAT. The consequences of DAT positivity are not well known and may point to early, asymptomatic disease, or to another disease associated with formation of RBC autoantibodies, such as a malignancy or (systemic) autoimmune disease. Currently, there are no guidelines to follow-up DAT positive donors.

A second unsolved difficulty is the choice of treatment in AIHA. Hemolysis can be stopped or at least attenuated with corticosteroids, aiming to inhibit autoantibody production and/or RBC destruction. Many patients do not respond adequately to corticosteroid treatment or develop severe side effects.

Currently, it is advised to avoid RBC transfusions since these may lead to aggravation of hemolysis and RBC alloantibody formation. But in case symptomatic anemia occurs, RBC transfusions need to be given. An evidence-based transfusion strategy for AIHA patients is needed to warrant safe transfusion in this complex patient group.

To design optimal diagnostic testing and (supportive) treatment algorithms, the investigators will study a group well-characterized patients with AIHA and blood donors without AIHA, via a prospective centralized clinical data collection and evaluation of new laboratory tests. With this data the knowledge of the AIHA pathophysiology and to evaluate diagnostic testing in correlation with clinical features and treatment outcome can be improved.

ELIGIBILITY:
Inclusion Criteria:

* Sufficient comprehension of the Dutch language
* Signed informed consent by patient and/or parent/caretaker or donor
* Patients older than 3 months
* Patients with a positive DAT, a positive eluate and signs of hemolysis*
* Patients with a positive DAT with complement only, negative eluate, but with signs of hemolysis
* Donors with a (repeatedly) positive DAT and a positive eluate and/or clinically relevant cold auto-antibodies

Exclusion Criteria:

* Prior inclusion in the DRAIHA study

Min Age: 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients, from the age of 3 months, with a positive DAT a positive eluate and signs of hemolysis and patients with a positive DAT for complement only with a negative eluate but with signs of hemolysis, and blood donors with a positive DAT and a positive eluate and/or clinically relevant cold autoantibodies.
Sampling Method: Non-Probability Sample
Enrollment: 720 (Estimated)
Dates: Start 2019-07-12 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Immunological characteristics of autoantibodies in autoimmune hemolytic anemia (AIHA) patients - laboratory tests. | 12-18 months
  Documentation of characteristics of autoantibodies (e.g. isotype, subtype, titer, thermal amplitude).
Assessment of hemolysis before and after therapy, reported per class of auto-immune hemolytic anemia. - laboratory tests | 12-18 months
  Documentation of hemolysis parameters (hemoglobin level (g/dL), reticulocytes (%), haptoglobin (mg/dL), bilirubin (μmol/L) and LDH(U/L)) before and after each type of therapy. AIHA classification as IgG/IgA only, IgG/IgA with complement activation or complement activation only.

SECONDARY OUTCOMES:
Incidence of underlying disease that causes or is associated with AIHA. | 12-18 months
  Documentation of physician-reported underlying disease that caused AIHA (e.g. autoimmune and/or lymphoproliferative disease, infection, medication).
Type of treatment prescribed as first-line, second-line or further-line treatment for AIHA. | 12-18 months
  The percentage of patients receiving first, second or further-line treatment for AIHA will be calculated.
Hematological response after each treatment line (CR, CR-u, PR and NR) | 12-18 months
  Percentage of patients with CR, CR-u, PR and NR after each treatment line. Hematological response will be classified as CR (complete remission), CR-u (CR- undetermined), PR (partial response) and NR (no response).
  CR: normal hemoglobin, no signs of hemolysis (normal haptoglobin, normal amount of reticulocytes, bilirubin, LDH), no treatment and transfusion independence during the last 4 weeks.
  CR-u: as CR, but hemoglobin, reticulocytes, LDH and/or bilirubin are deviating through another reason (e.g. underlying malignant disease).
  PR: 1. Hemoglobin > 10g/dL, no signs of hemolysis, transfusion independent, but a continuous treatment with low dose prednisone (< 10 mg/day) or other immunosuppressive therapy is necessary. 2. Compensated hemolytic anemia with an stable hemoglobin >10g/dL, transfusion independent, maximal dose of prednisone < 10mg/day or other continuous immunosuppressive therapy or EPO.
  NR: no PR reached
Relapse-free survival, defined as the time since the achievement of complete or partial remission until relapse of AIHA or dead from any cause. | 12-18 month
  Relapse-free survival will be calculated as the time since the achievement of complete or partial remission until relapse of AIHA or dead from any cause. Median RFS and 95% CI will be calculated.
Documentation of adverse events during the treatment of AIHA. | 12-18 month
  Documentation of adverse events during the treatment of AIHA indicated according to the Common Terminology Criteria for Adverse Events v4.0 (CTCAE) Publish Date: May 28, 2009
Assessment of hemolysis parameters after red blood cell transfusion. | 1 and 7 days after transfusion
  Documentation of hemolysis parameters (hemoglobin level (g/dL), reticulocytes (%), haptoglobin (mg/dL), bilirubin (μmol/L) and LDH (U/L)) before red blood cell transfusion.
Change in the incidence of auto- and alloantibodies after red blood cell transfusion. | 12-18 months
  Compare the incidence of auto- and alloantibodies before and after red blood cell transfusion.
Characteristics of autoantibodies of DAT positive blood donors. | 12-18 months
  Documentation of characteristics of autoantibodies (e.g. isotype, subtype, titer, thermal amplitude) of DAT positive blood donors.

CONTACTS AND LOCATIONS:
Overall Officials: M. De Haas, Prof. MD PhD, Principal Investigator — Center for Clinical Transfusion Research (CCTR), Sanquin, The Netherlands; S.S Zeerleder, Prof. MD PhD, Principal Investigator — University Hospital, University of Bern, Switzerland and Department for BioMedical Research, University of Bern, Switzerland
Locations (2):
- Netherlands (2):
  - AMC, Amsterdam-Zuidoost
  - UMC Radboud, Nijmegen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garratty G. Immune hemolytic anemia associated with negative routine serology. Semin Hematol. 2005 Jul;42(3):156-64. doi: 10.1053/j.seminhematol.2005.04.005. PMID 16041665
- [Background] Freedman J. False-positive antiglobulin tests in healthy subjects and in hospital patients. J Clin Pathol. 1979 Oct;32(10):1014-8. doi: 10.1136/jcp.32.10.1014. PMID 521494
- [Background] Barcellini W, Fattizzo B, Zaninoni A, Radice T, Nichele I, Di Bona E, Lunghi M, Tassinari C, Alfinito F, Ferrari A, Leporace AP, Niscola P, Carpenedo M, Boschetti C, Revelli N, Villa MA, Consonni D, Scaramucci L, De Fabritiis P, Tagariello G, Gaidano G, Rodeghiero F, Cortelezzi A, Zanella A. Clinical heterogeneity and predictors of outcome in primary autoimmune hemolytic anemia: a GIMEMA study of 308 patients. Blood. 2014 Nov 6;124(19):2930-6. doi: 10.1182/blood-2014-06-583021. Epub 2014 Sep 16. PMID 25232059
- [Background] Rottenberg Y, Yahalom V, Shinar E, Barchana M, Adler B, Paltiel O. Blood donors with positive direct antiglobulin tests are at increased risk for cancer. Transfusion. 2009 May;49(5):838-42. doi: 10.1111/j.1537-2995.2008.02054.x. Epub 2009 Jan 2. PMID 19170992
- [Background] Meulenbroek EM, de Haas M, Brouwer C, Folman C, Zeerleder SS, Wouters D. Complement deposition in autoimmune hemolytic anemia is a footprint for difficult-to-detect IgM autoantibodies. Haematologica. 2015 Nov;100(11):1407-14. doi: 10.3324/haematol.2015.128991. Epub 2015 Sep 9. PMID 26354757
- [Background] Zanella A, Barcellini W. Treatment of autoimmune hemolytic anemias. Haematologica. 2014 Oct;99(10):1547-54. doi: 10.3324/haematol.2014.114561. PMID 25271314
- [Background] Reynaud Q, Durieu I, Dutertre M, Ledochowski S, Durupt S, Michallet AS, Vital-Durand D, Lega JC. Efficacy and safety of rituximab in auto-immune hemolytic anemia: A meta-analysis of 21 studies. Autoimmun Rev. 2015 Apr;14(4):304-13. doi: 10.1016/j.autrev.2014.11.014. Epub 2014 Dec 9. PMID 25497766
- [Background] Shi J, Rose EL, Singh A, Hussain S, Stagliano NE, Parry GC, Panicker S. TNT003, an inhibitor of the serine protease C1s, prevents complement activation induced by cold agglutinins. Blood. 2014 Jun 26;123(26):4015-22. doi: 10.1182/blood-2014-02-556027. Epub 2014 Apr 2. PMID 24695853
- [Background] Wouters D, Stephan F, Strengers P, de Haas M, Brouwer C, Hagenbeek A, van Oers MH, Zeerleder S. C1-esterase inhibitor concentrate rescues erythrocytes from complement-mediated destruction in autoimmune hemolytic anemia. Blood. 2013 Feb 14;121(7):1242-4. doi: 10.1182/blood-2012-11-467209. No abstract available. PMID 23411737